CLINICAL TRIAL: NCT00844103
Title: A Phase I, Randomised, Double Blind, Placebo-Controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of Multiple Oral Doses of AZD8566 in Healthy Volunteers
Brief Title: Study to Investigate the Safety, Tolerability and Pharmacokinetics of Multiple Doses of AZD8566.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Harsukh Parmar , Medical Science Director, Respiratory and Inflammation Emerging Product Team, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D1320C00002
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2009-04-30 (Estimated); Status verified 2009-04

CONDITIONS: Pharmacokinetics
Keywords: Volunteer; Safety; Tolerability; AZD8566

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD8566
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8566 — 10ml oral solution administered once a day over 10 days. Specific dose will be selected by the safety review committee
  Arms: 1
Drug: Placebo — 10ml oral solution administered once a day over 10 days.
  Arms: 2

SUMMARY:
The purpose of this study is to determine how well tolerated and safe AZD8566 is when given over 10 days, at different dose levels. This study will also determine how AZD8566 is distributed around the body and how it leaves the body.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent.
* Clinically normal physical findings and laboratory values as judged by the investigator with normal ECG
* Females who are permanently or surgically sterile or postmenopausal and males.

Exclusion Criteria:

* Intake of medicine (except Hormone Replacement Therapy or occasional paracetamol) within 3 weeks before first administration of study drug
* History of any convulsions or seizures
* History of infection or at risk of infection due to recent surgery or trauma
* History or presence of conditions known to interfere with the absorption, distribution, metabolism and excretion of the study drug

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile: concentration of AZD8566 in blood | Samples taken during Visit 2 (residential period) at up to 15 defined timepoints pre-dose and post- dose on Day 1 and Day 10
Safety and tolerability of AZD8566 by assessment of vital signs, laboratory variables, ECG and adverse events | Assessments taken at Visit 1 (enrolment), defined timepoints pre-dose and post-dose during Visit 2 (residential period) and at Visit 3 (follow up). Volunteers will be monitored throughout the study from Visit 1 to Visit 3 for adverse events.

SECONDARY OUTCOMES:
Pharmacokinetic profile: concentration of AZD8566 in urine | Samples collected over 48 hours from pre-dose to 48 hours post-dose on Day 1 and Day 10.

CONTACTS AND LOCATIONS:
Overall Officials: Emeline Ramos, MD, Principal Investigator — Clinical Pharmacology Unit
Locations (1):
- Research Site, Macclesfield, Cheshire, United Kingdom